CLINICAL TRIAL: NCT02066012
Title: Impact of Dysmetabolic Iron Overload Syndrome on Polarization Capacity of Macrophages
Brief Title: MEPHISTO (Macrophage Phenotype In Metabolic Syndrome With Iron Overload)
Acronym: MEPHISTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0180; 2013-A01687-38
Record Dates: First submitted 2014-02-14; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Dysmetabolic Iron Overload Syndrome; Metabolic Syndrome X
Keywords: Dysmetabolic Iron Overload Syndrome; Metabolic Syndrome X; Iron; Monocyte; Macrophage; Polarization
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- group DIOS: group DIOS composed of subjects with dysmetabolic hepatosiderosis
  Interventions: Other: dysmetabolic iron overload syndrome
- group M: group M composed of subjects with metabolic syndrom without iron overload
  Interventions: Other: dysmetabolic iron overload syndrome
- group T: group T composed of lean subjects
  Interventions: Other: dysmetabolic iron overload syndrome

INTERVENTIONS:
Other: dysmetabolic iron overload syndrome

SUMMARY:
Dysmetabolic iron overload syndrome (DIOS), is a frequent hepatic iron overload associated with metabolic syndrome. We hypothesize that this mild iron overload can induce a increased macrophagic polarization towards inflammatory types, thereby contributing to cardiovascular risk. Our main objective is to highlight the influence of iron overload on polarization capacity of monocytes into alternative macrophages (called M2). We therefore compare phenotypic markers of monocytes/macrophages between subjects with DIOS, metabolic syndrome without iron overload and lean subjects.

DETAILED DESCRIPTION:
MEPHISTO is a pathophysiological, transverse, case-control, single-center study (university hospital, Clermont-Ferrand, France). No intervention (drug or nutritional) is conducted as part of this study and the participants are not subject to any exclusion period. Our objective is to investigate the effects of iron overload on monocyte/macrophage polarization and its relations with the cardiovascular risk factors.

We study 60 subjects divided into 3 groups of 20 participants :

* group DIOS composed of subjects with dysmetabolic hepatosiderosis
* group M composed of subjects with metabolic syndrom without iron overload
* group T composed of lean subjects DIOS group participants were selected among patients recently diagnosed as DIOS, without any secondary hyperferritinemia and with hepatic iron overload proved by liver MRI.

Recruitement of group DIOS was carried out in the internal medicine service. Subjects of group M and DIOS come from the file of volunteers from the center of clinical investigation (CIC-501, Clermont-Ferrand). Subject of group M to group DIOS are matched by age, gender (+/- 5 kg/m²) and BMI. Subjects of group T to group DIOS are matched by age and gender. As no direct benefit is expected for the participants, they receive a lump sum compensation of 50 euros.

Each participant undergoes only a 1 hour consultation including a clinical examination and blood sample.

We focus on clinical parameters of the metabolic syndrome (waist size, BMI, blood pressure) and on seeking exclusion factors (infection, neoplasia, anti-inflammatory drugs). Due to their potential influence on inflammation and oxidant stress, these factors, as same as smoking were excluded.

Blood sample will be used to perform:

* classical laboratory test (blood count, reticulocytes, ASAT, ALAT, LDH, lipid profile, glycemia, insulinemia, TSH, , vitamin D, ferritin, transferrin saturation, CRP),
* specific dosages (IL-6, TNFalpha, hepcidine) by ELISA,
* monocyte phenotype ( CD14, CD16, CD 163, MR) by FACS (Fluorescence Activated Cell Sorting),
* measurement of the gene expression from monocytes and macrophages after culturing by real-time PCR.

Our main analysis focus on ex vivo polarization of monocytes into alternative macrophages (M2) and phenotypic characterization. Before and after culturing monocytes with (to induce M2 macrophage) or without IL-4 (to induce resident macrophage), we will measure the expression of phenotypic markers of polarization (MR, CD200R, F13A1, CD163, AMAC1, TGFb), inflammatory markers (TNFα , MCP- 1, IL-6) , oxidative stress markers (HO- 1 ), and markers of iron metabolism (ferroportin, ferritin, hepcidin). We use quantitative PCR microfluidic card (TLDA, Taqman Low-Density Array) to measure gene expression of monocytes and type M2 macrophages. This technique allows screening of expression for 24 genes. Different phases are required: RNA extraction (RNeasy kit, Qiagen), the reverse transcription (RT-PCR kit, HighCap cDNA RT kit, Applied Biosystems), amplification (TaqMan Fast Advanced Master Mix, Applied Biosystems), and finally the study of gene expression (MFC TaqMan Array for GeneEx, Format 24, Applied Biosystems). Our main outcome is capacity of polarization in M2 macrophages evidenced by expression of MR, CD200R, F13A1, CD163, AMAC1, TGFb. Evaluating the influence of iron overload on data from the clinical examination, the results of standard biology and monocyte gene expression is our secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* • 18 years old and over

  * written consent
  * for groups M and HSD at least one criteria of the metabolic syndrome definition according to the International Diabetes Federation
  * for group M only hepatic iron overload mesured by IRM (above 50 µmol/g) hyperferritnemia between 450 and 1500 µg/l
  * for group T only BMI < 25 kg/m² Waist size < 80 cm for women and <94 cm for men

Exclusion Criteria:

* persons under guardianship
* pregnancy
* active smoking
* current inflammatory or cancerous disease
* hereditary hemochromatosis
* use of anti-inflammatory, immunosuppressive or hypoglycaemic drugs
* hemolysis
* alcool consumption above 14 doses for women and 21 doses for men per week
* history of therapeutic phlebotomy
* inflammatory syndrome with CRP above 15 mg/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: metabolic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Expression (RNA) of macrophagic polarization markers | at day 1
  Expression (RNA) of macrophagic polarization markers (MR, CD200R, F13A1, CD163, AMAC1, TGFβ), among subjects with or without iron overload

SECONDARY OUTCOMES:
characteristics of the subjects | at day 1
  Statistical relationships between monocyte phenotype and clinical (metabolic abnormalities) or biological (level of iron overload, oxidative stress and insulino-resistance) characteristics of the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Marc RUIVARD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France